CLINICAL TRIAL: NCT07178951
Title: Safety and Feasibility of the Neurolyser XR Device for the Treatment of Predominantly Medial Chronic Knee Pain Due to Osteoarthritis
Brief Title: Neurolysis for the Treatment of Medial Chronic Knee Pain Due to Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: FUSMobile Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Knee-001
Record Dates: First submitted 2025-06-15; First posted 2025-09-17 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis (OA) of the Knee; Knee Pain Arthritis; Chronic Knee Pain
Keywords: osteoarthritis; knee pain; focused ultrasound; nerve ablation
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: pilot, single center, prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thermal ablation with Neurolyser XR (Experimental): Ablation of sensory nerves in the knee joint
  Interventions: Device: Neurotomy of the medial sensory articular branches

INTERVENTIONS:
Device: Neurotomy of the medial sensory articular branches — Non-invasive thermal ablation of the medial sensory articular branches of the knee joint
  Other Names: Nerve ablation; genicular nerve ablation

SUMMARY:
This study involves the use of sound waves to block pain signals caused by osteoarthritis of the knee. The sound waves are tightly focused on a specific area of the nerve. The sound waves cause a break in the nerve which carries pain signals. Sound waves transmit through the skin so there is no need for needles. The procedure takes approximately one hour. The device has been approved in Health Canada and Europe for the treatment of lower back pain. This study is to evaluate the use of the same device for people in Canada who have knee pain related to osteoarthritis.

DETAILED DESCRIPTION:
The research staff will provide a detailed description of the procedure to the study participant live, allowing time for the participant to ask questions. Once the participant agrees to be in the study, an informed consent form will be signed.

Throughout the study, the research team will closely follow the participants health as it is related to their knee. The participant will have a physical exam of their knee and a pressure algometry test at each onsite visit. They will also rate their pain level on a numerical scale, provide a history of medications taken, and complete several quality of life questionnaires.

The participant will be asked to take their usual pain medication prior to the procedure. The study doctor may also provide additional medication depending on the study participants situation.

The study procedure will last approximately 1 hour. The procedure will take place using a standard X-ray device which allows the study doctor to see the structure of the knee and allow for location of the nerve causing knee pain.

The study device will use ultrasound waves to cause damage to the nerve of the knee where the pain is generated. The goal is to interrupt the pain signal pathway. The ultrasound waves go through the skin so no needles or incisions are needed.

It is unknown how much pain relief the participant will feel or how long it will last. The purpose of the study is to evaluate ten people who have the study procedure. If the study results are good, the manufacturer of the device plans to open up a larger study to involve more study participants.

For participants who have access and a MRI is not contraindicated, a follow-up MRI exam will be performed from day 5 to 7 of the participant's knee.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate to severe, predominantly medial chronic knee pain
2. Age adult >18 years old
3. WOMAC Score of 30 or higher
4. NRS>6 with ambulation
5. Radiological confirmation of knee osteoarthritis (Kellgren-Lawrence Scale: 2-4)
6. Participants in whom the measured skin to bone depth is 2-6 cm using imaging ultrasound and ultrasound gel pad in the upper medial and lower medial joint capsule targets.

Exclusion Criteria:

1. Individuals meeting any of the following criteria are not eligible for participation in this study:
2. Individuals after any surgery associated with altered integrity of bone structure
3. Individuals with severe pain in the second knee
4. Individuals unable to understand and complete the research questionnaires in the official language
5. Individuals presenting with any severe medical condition preventing the participant from safely and effectively being treated in the study or reporting study outcomes, per PI decision
6. Individuals with extensive scarring of the skin and tissue overlying the treatment area
7. Individuals enrolled in or planned to be enrolled in another clinical trial during the duration of this research project
8. Individuals with active inflammatory (e.g., rheumatoid) arthritis
9. Individuals with concomitant mental health disorders, excluding compensated mood disorders
10. Individuals with altered perception and processing of pain: Average NRS > 9, PCS>30, SSS-8 > 11, CSI>40 [46], [47], [48]
11. Individuals with a first-degree family member already enrolled in this study
12. Individuals who are scheduled for any interventional/surgical procedure within 3 months from the screening date, excluding trivial surgeries (e.g., cataract, skin tumors)
13. Inability to attend follow-up visits and physiotherapy due to travel distance or other restrictions
14. Symptomatic multifocal nociplastic chronic pain (e.g., fibromyalgia, generalized osteoarthritis) or any other chronic pain condition that could influence symptoms.
15. Participants who have undergone radiofrequency ablation of the genicular nerves in the planned treatment limb within the preceding 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
A positive clinical outcome will be measured by a 2-point reduction in the Numerical Rating Score (NRS) | Baseline score will be compared to post procedure intervals at 2 days, 7 days, 1 month, 3 months, and 6 months.
  The NRS score is a 10 point scale, 0 to 10, with 0 meaning "no pain" and 10 meaning "worst possible pain"; the NRS score will be measured at baseline and all follow-up intervals - 2 days, 7 days, 1 month, 3 months, and 6 months..
Safety will be measured by the incidence and severity of treatment-related adverse events. | Adverse events will be evaluated at baseline and post procedure - 2 days, 7 days, 1 month, 3 months, and 6 months.
  Adverse events will be evaluated throughout the study.

SECONDARY OUTCOMES:
Lesion size and location | Participants will have an MRI 5-7 days post treatment when feasible and not contraindicated
  Lesion size and location as shown in MRI images post treatment as available
Procedure time (in minutes) | The time of the procedure will be documented in minutes.
  Procedure time will be documented from start to finish
Radiation exposure (in seconds) | The fluoroscopy time will be calculated and documented during the procedure.
  The procedure is completed using fluroscopy. The fluroscopy time is calculated by the C-Arm. This number will be documented.
Periprocedural analgesic/sedative requirement | During the procedure, analgesic/sedative use will be documented.
  Analgesic/sedatives used during the procedure will be documented.
Change in Pain Pressure Threshold (PPT) as measured on the tibial plateau. | The PPT will be evaluated and documented at baseline and at follow-up intervals - 2 days, 7 days, 1 month, 3 months, and 6 months
  A pressure algometry device will be used to measure the pain pressure threshold throughout the study.
Change in score Patient Global Impression of Change (PGIC) | PGIC questionnaires will be provided to participants 1 month, 3 months, and 6 months post procedure.
  The PGIC questionnaire will be given to participants during their onsite follow up visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Unika Medical Centre, North York, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
This is a pilot study. If results are positive, we plan to organize a larger pivotal study.